CLINICAL TRIAL: NCT02728063
Title: Effect of a Mixture of Probiotics, Lactibiane Tolérance® on Intestinal Permeability in Individuals Suffering From Irritable Bowel Syndrome With Diarrheal Predominance
Brief Title: Lactibiane Tolérance® in Individuals Suffering From Irritable Bowel Syndrome With Diarrheal Predominance
Acronym: PILATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PiLeJe (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PEC15144
Record Dates: First submitted 2016-03-08; First posted 2016-04-05 (Estimated); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Diarrhea Predominant Irritable Bowel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm (Experimental): Supplementation with Lactibiane Tolerance
  Interventions: Dietary Supplement: Lactibiane Tolerance

INTERVENTIONS:
Dietary Supplement: Lactibiane Tolerance — probiotics

SUMMARY:
The main objective of the study is to evaluate the effect on intestinal permeability of a supplementation with Lactibiane Tolérance® for 4 weeks (28 days) in patients suffering from irritable bowel syndrome (IBS) with diarrhea predominance.

Secondary objectives of the study are to evaluate the effects of supplementation with Lactibiane Tolérance® for 4 weeks (28 days) in patients suffering from IBS with diarrhea predominance on intestinal permeability, inflammation of the digestive tract, symptoms and comfort.

Single-center study in single open arms: 30 volunteer adults suffering from Irritable Bowel Syndrome (IBS) with diarrhea predominance and matching the criteria of inclusion and non-inclusion listed below.

DETAILED DESCRIPTION:
single-center pilot study in single open arm:

* 2 to 6 weeks before enrollment: a screening visit (visit 0 [V0]) is carried out for verification of eligibility. time between V0 and V1 is a wash-out period with a duration decided by the physician (max 8 weeks).
* The experimental phase is composed of 2 visits (Visit 1 [V1] and Visit 2 [V2]) separated by 28 days (± 2 days) : from V1 to V2 patients are taking the product Lactibiane Tolérance®.
* V1 and V2 each include collection of stools, a blood sample, questionnaires on abdominal symptoms and quality of life, dynamic test of absorption of lactulose / mannitol to evaluate the intestinal permeability, recto-sigmoidoscopy with confocal endomicroscopy for in-vivo study of fluorescein leakage in the lamina propria and biopsies for ex-vivo measurements.
* "carmine red" test for the evaluation of intestinal transit speed is carried out the week before V1 and V2 (at least 72 hours before the visit). Questionnaires on abdominal symptoms as well as the frequency and consistency of stools are filled during the 7 days before V1 and V2 before.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 75;
* With symptoms of IBS with predominant diarrhea according to the Rome III criteria;
* For women of childbearing age: effective contraception and agreement to keep it throughout the study;
* General and mental health compatible with participation in the study and to be followed as an outpatient in the opinion of the investigator: no clinically significant and relevant abnormality according to medical history and physical examination;
* Agreeing to maintain their lifestyle during the study (same eating habits and physical activity);
* Able and willing to participate in research in accordance with the protocol procedures particularly regarding consumption of the product under consideration and having signed an informed consent form dated;
* Belonging to a social security scheme;
* Willing to be included in the file of volunteers participating in biomedical research.

Exclusion Criteria:

* Having a history of hypersensitivity to any of the ingredients of the product under consideration;
* Having a history of hypersensitivity to fluorescein and / or red carmine (E120 food coloring);
* With immunodeficiency or with a severe or progressive disease (cardiac, pulmonary, hepatic, renal, hematologic, neoplastic, or infectious);
* With acute or severe chronic disease (chronic alcoholism, drug addiction) found incompatible with participation in the study by the investigator;
* Suffering from a metabolic disorder or a chronic inflammatory digestive disease affecting the intestinal transit or absorption of nutrients such as diabetes, hyperthyroidism, celiac disease or Crohn's disease;
* Having a medical history or current condition that, according to the investigator, may interfere with the results of the study or expose the subject to additional risk;
* Currently under medication or food supplement treatment, according to the investigator, may interfere with the results of the study or stopped within too short before inclusion in V1 (less than a month for antibiotics, pre and probiotics, less than 14 days for antidiarrheal, steroidal anti-inflammatories, NSAIDs, aspirin, antihistamines and drugs. treatment with maximum 2 concomitant psychotropic can be tolerated only if it exists for more than 3 months before inclusion);
* Having a lifestyle incompatible with the study by the investigator;
* Woman during pregnancy or breastfeeding or planning to become pregnant within 2 months;
* Planning to travel and hold during the study period or impossible to contact in case of emergency;
* Having a psychological or linguistic inability to understand and sign the informed consent;
* Participating in another clinical trial or exclusion period of a previous clinical trial;
* Having received over the past 12 months, no more than 4,500 euros in payment for participation in clinical trials;
* Under legal protection (guardianship, trusteeship) or deprived of his rights under the administrative or judicial decision.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-05-11 (Actual); Primary Completion 2018-04-11 (Actual); Study Completion 2018-04-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline of intestinal permeability | at day 0 and day 28
  Evolution between V1 and V2 of intestinal permeability evaluated by the lactulose-mannitol test according to the slope of urinary excretion of ingested lactulose percentage (calculated by linear regression) during the period representing the passage into the small intestine (2 to 4 hours after ingestion of lactulose-mannitol mixture).

SECONDARY OUTCOMES:
Change from baseline of intestinal permeability - secondary 1 | at day 0 and day 28
  Evolution of slope percentages urinary excretion (UE) of ingested mannitol ([M]) (calculated by linear regression) during the period representing the Passage Into the Small Intestine (PISI) (2 to 4 hours (h) after ingestion of [L]-[M] mixture)
Change from baseline of intestinal permeability - secondary 2 | at day 0 and day 28
  Evolution of the ratio between the slopes of the UE percentages of lactulose ([L]) and [M] ingested during the PISI (2 to 4h after ingestion of lactulose-mannitol mixture)
Change from baseline of intestinal permeability - secondary 3 | at day 0 and day 28
  Evolution of the percentage of UE of [L] ingested on the excretion of ingested [M] during the period representing the PISI (2 to 4h after ingestion)
Change from baseline of intestinal permeability - secondary 4 | at day 0 and day 28
  Evolution of the UE percentage of [L] ingested on the UE of ingested [M] each lap of the period representing the PISI
Change from baseline of intestinal permeability - secondary 5 | at day 0 and day 28
  Evolution of he percent UE of [L] ingested on the UE of ingested [M] during the period representing the passage in the colon (between 4 and 5h after ingestion)
Change from baseline of intestinal permeability - secondary 6 | at day 0 and day 28
  Evolution of the percent UE of [L] ingested on the UE of ingested [M] during the period of 5h after ingestion
Change from baseline of intestinal permeability - secondary 7 | at day 0 and day 28
  Evolution of the UE percentage of [L] ingested on the UE of ingested [M] during the transition period representative of the stomach to the small intestine (between 0 and 2h after
Change from baseline of intestinal permeability - secondary 8 | at day 0 and day 28
  Evolution of the Percentage of UE of [L] and [M] ingested during the period representing the PISI (2 to 4h after ingestion)
Change from baseline of intestinal permeability - secondary 9 | at day 0 and day 28
  Evolution of the Percentage of UE of [L] and [M] ingested during a period of 5h after ingestion
Change from baseline of intestinal permeability - secondary 10 | at day 0 and day 28
  Evolution of the Percentage of UE of [L] and [M] ingested each 5h lap
Change from the baseline of the inflammatory status - secondary 11 | at day 0 and day 28
  Evolution between V1 and V2 of inflammatory status by fecal calprotectin
Change from the baseline of the symptomatology - secondary 12 | at week 0 and week 4
  Time to onset of the first colored red stool after taking carmine red capsules (minutes)
Change from the baseline of the symptomatology - secondary 13 | at week 0 and week 4
  Average intensity of 7 days of the worst abdominal pain on Likert scale (11 points)
Change from the baseline of the symptomatology - secondary 14 | at week 0 and week 4
  Medium intensity of 7 days of abdominal discomfort on Likert scale (11 points)
Change from the baseline of the symptomatology - secondary 15 | at week 0 and week 4
  Stool consistency average of 7 days after Bristol Stool Scale (BSS)
Change from the baseline of the symptomatology - secondary 16 | at week 0 and week 4
  Mean daily stool frequency of 7 days after BSS quiz

OTHER OUTCOMES:
Parameters measured ex vivo from colonic biopsies placed in Ussing chamber : change from baseline of paracellular permeability | at day 0 and day 28
  Evolution of the slope ( determined by linear regression ) and area under the curve of evolution of the concentration of sulfonic acid fluorescence (measured in the basolateral chamber ) over time (measured every 30 min for 3 hours )
Parameters measured ex vivo from colonic biopsies placed in Ussing : change from baseline of transcellular permeability | at day 0 and day 28
  Evolution of the slope ( calculated by linear regression) and area under the curve of evolution of the concentration of Horse Radish Peroxidase (HRP) (measured in the basolateral chamber ) over time (measured every 30 minutes between 1 and 3 hours) .

CONTACTS AND LOCATIONS:
Overall Officials: Coron Emmanuel, Pr., Principal Investigator — Nantes University Hospital
Locations (1):
- CHU-Hôtel-Dieu, Service d'Hépato-gastro-entérologie, Nantes, France

IPD SHARING:
Plan to Share IPD: No